CLINICAL TRIAL: NCT05822830
Title: A Phase 3b, Randomized Controlled Study to Evaluate the Efficacy and Safety of Tirzepatide Compared to Semaglutide in Adults Who Have Obesity or Overweight With Weight Related Comorbidities
Brief Title: A Study of Tirzepatide (LY3298176) in Participants With Obesity or Overweight With Weight Related Comorbidities
Acronym: SURMOUNT-5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17203; I8F-MC-GPHJ (Other: Eli Lilly and Company); U1111-1283-5404 (Other: UTN Number)
Record Dates: First submitted 2022-09-16; First posted 2023-04-21 (Actual); Results first posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Obesity; Overweight
Keywords: Metabolism and Nutrition; Disorder; Prediabetes; Diet; Exercise
MeSH Terms: conditions — Obesity; Overweight; Disease; Prediabetic State; Motor Activity | interventions — Tirzepatide; semaglutide

STUDY DESIGN:
Intervention Model Description: Phase 3b
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 15 mg or MTD - Tirzepatide (Experimental): Participants received a starting dose of 2.5 milligrams (mg) tirzepatide administered subcutaneously (SC) once weekly (QW) for 4 weeks, then the dose was increased by 2.5 mg every 4 weeks (2.5 to 5 to 7.5 to 10 to 12.5 to 15 mg) up to 15 mg QW or maximum tolerated dose [MTD (10 mg or 15 mg)] until Week 72.
  Interventions: Drug: Tirzepatide
- 2.4 mg or MTD - Semaglutide (Active Comparator): Participants received a starting dose of 0.25 mg semaglutide administered SC QW for 4 weeks, then the dose was increased every 4 weeks (0.25 to 0.5 to 1.0 to 1.7 to 2.4 mg) up to 2.4 mg QW or MTD (1.7 mg or 2.4 mg) until Week 72.
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: 15 mg or MTD - Tirzepatide
Drug: Semaglutide — Administered SC
  Arms: 2.4 mg or MTD - Semaglutide

SUMMARY:
The main purpose of this phase 3b study is to evaluate the efficacy and safety of tirzepatide compared with semaglutide in adult participants who have obesity or overweight with weight related comorbidities without Type 2 Diabetes. The study will last around 74 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) of ≥30 kilogram per square meter (kg/m²) or ≥27 kg/m² and previously diagnosed with at least one of the following weight related comorbidities: hypertension, dyslipidemia, obstructive sleep apnea, cardiovascular disease
* Have a history of at least 1 unsuccessful dietary effort to lose body weight

Exclusion Criteria:

* Diabetes mellitus
* Change in body weight greater than 5 kg within 3 months prior to starting study
* Obesity induced by other endocrinologic disorders or monogenetic or syndromic forms of obesity
* History of pancreatitis
* Family or personal history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN-2)
* History of significant active or unstable major depressive disorder (MDD) or other severe psychiatric disorder within the last 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 751 (Actual)
Dates: Start 2023-04-21 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2024-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (32):
- United States (30):
  - Cahaba Research, Birmingham, Alabama
  - Cahaba Research - Pelham, Pelham, Alabama
  - Southern California Dermatology, Inc., Santa Ana, California
  - Encompass Clinical Research, Spring Valley, California
  - University Clinical Investigators, Inc., Tustin, California
  - Velocity Clinical Research, Hallandale Beach, Hallandale, Florida
  - New Horizon Research Center, Miami, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Rophe Adult and Pediatric Medicine/SKYCRNG, Union City, Georgia
  - Rocky Mountain Clinical Research, Idaho Falls, Idaho
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - L-MARC Research Center, Louisville, Kentucky
  - Arcturus Healthcare , PLC, Troy Internal Medicine Research Division, Troy, Michigan
  - Prime Health and Wellness/SKYCRNG, Fayette, Mississippi
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Palm Research Center Tenaya, Las Vegas, Nevada
  - Palm Research Center Sunset, Las Vegas, Nevada
  - Weill Cornell Medical College, New York, New York
  - PharmQuest, Greensboro, North Carolina
  - Lillestol Research, Fargo, North Dakota
  - Alliance for Multispecialty Research, LLC, Norman, Oklahoma
  - Tribe Clinical Research, LLC, Greenville, South Carolina
  - WR-Clinsearch, LLC, Chattanooga, Tennessee
  - The University of Texas Health Science Center at Houston, Bellaire, Texas
  - Dallas Diabetes Research Center, Dallas, Texas
  - North Texas Endocrine Center, Dallas, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - PlanIt Research, PLLC, Houston, Texas
  - Southern Endocrinology Associates, Mesquite, Texas
  - Pinnacle Clinical Research, San Antonio, Texas
- Puerto Rico (2):
  - Puerto Rico Medical Research, Ponce
  - Wellness clinical Research Vega Baja, Vega Baja

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org

REFERENCES:
- [Derived] Mamas MA, Bays H, Li R, Upadhyay N, Irani T, Senyucel C, Dunn JP, Liu-Seifert H. Tirzepatide compared with semaglutide and 10-year cardiovascular disease risk reduction in obesity: post-hoc analysis of the SURMOUNT-5 trial. Eur Heart J Open. 2025 Sep 2;5(5):oeaf117. doi: 10.1093/ehjopen/oeaf117. eCollection 2025 Sep. PMID 40980721
- [Derived] Aronne LJ, Horn DB, le Roux CW, Ho W, Falcon BL, Gomez Valderas E, Das S, Lee CJ, Glass LC, Senyucel C, Dunn JP; SURMOUNT-5 Trial Investigators. Tirzepatide as Compared with Semaglutide for the Treatment of Obesity. N Engl J Med. 2025 Jul 3;393(1):26-36. doi: 10.1056/NEJMoa2416394. Epub 2025 May 11. PMID 40353578
- See also: A Study of Tirzepatide (LY3298176) in Participants With Obesity or Overweight With Weight Related Comorbidities (SURMOUNT-5) — https://trials.lilly.com/en-US/trial/399775

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 15 mg or MTD - Tirzepatide | 2.4 mg or MTD - Semaglutide
Started | 375 | 376
Received At Least One Dose of Study Drug | 374 | 376
Completed | 319 | 319
Not Completed | 56 | 57
Not completed — Adverse Event | 6 | 6
Not completed — Assigned Treatment by Mistake | 5 | 3
Not completed — Lost to Follow-up | 16 | 18
Not completed — Non-Compliance With Study Drug | 1 | 1
Not completed — Participant was Out of the Country | 0 | 1
Not completed — Pregnancy | 1 | 2
Not completed — Withdrawal by Subject | 27 | 26

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- 15 mg or MTD - Tirzepatide: Participants received a starting dose of 2.5 mg tirzepatide administered SC QW for 4 weeks, then the dose was increased by 2.5 mg every 4 weeks (2.5 to 5 to 7.5 to 10 to 12.5 to 15 mg) up to 15 mg QW or MTD (10 mg or 15 mg) until Week 72.
- Total: Total of all reporting groups
Arm/Group | 15 mg or MTD - Tirzepatide | 2.4 mg or MTD - Semaglutide | Total
Number analyzed (Participants) | 374 | 376 | 750
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.00 (12.94) | 44.40 (12.74) | 44.70 (12.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 242 | 243 | 485
  Male | 132 | 133 | 265
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 93 | 103 | 196
  Not Hispanic or Latino | 281 | 273 | 554
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 0 | 6
  Asian | 11 | 7 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 77 | 67 | 144
  White | 276 | 295 | 571
  More than one race | 4 | 7 | 11
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 374 | 376 | 750

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Body Weight
Description: Percent change from baseline in body weight was reported. Least Squares (LS) mean was determined using ANCOVA model with Baseline + Baseline BMI Group 1 + Sex + Pre diabetes status at randomization + Treatment (Type III sum of squares) as variables.
Time Frame: Baseline, Week 72
Population: All participants who received at least one dose of study drug and had evaluable data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | 15 mg or MTD - Tirzepatide | 2.4 mg or MTD - Semaglutide
Number analyzed (Participants) | 318 | 318
Percent change | -20.2 (0.59) | -13.7 (0.59)
Statistical Analysis 1: Comparison: 15 mg or MTD - Tirzepatide vs 2.4 mg or MTD - Semaglutide; Test type: Superiority; LS Mean Difference = -6.5, 95% CI 2-sided [-8.1 to -4.9]

2. Secondary Outcome: Percentage of Participants Who Achieve ≥10% Body Weight Reduction
Description: Percentage of participants who achieved ≥10% body weight reduction (observed values) was reported.
Time Frame: Week 72
Population: All participants who received at least one dose of study drug and had evaluable data for this outcome.
Measure: Number; unit: Percentage of participants
Arm/Group | 15 mg or MTD - Tirzepatide | 2.4 mg or MTD - Semaglutide
Number analyzed (Participants) | 318 | 318
Percentage of participants | 87.7 | 66.7

3. Secondary Outcome: Percentage of Participants Who Achieve ≥15% Body Weight Reduction
Description: Percentage of participants who achieved ≥15% body weight reduction (observed values) was reported.
Time Frame: Week 72
Population: All participants who received at least one dose of study drug and had evaluable data for this outcome.
Measure: Number; unit: Percentage of participants
Arm/Group | 15 mg or MTD - Tirzepatide | 2.4 mg or MTD - Semaglutide
Number analyzed (Participants) | 318 | 318
Percentage of participants | 71.7 | 45.0

4. Secondary Outcome: Percentage of Participants Who Achieve ≥20% Body Weight Reduction
Description: Percentage of participants who achieved ≥20% body weight reduction (observed values) was reported.
Time Frame: Week 72
Population: All participants who received at least one dose of study drug and had evaluable data for this outcome.
Measure: Number; unit: Percentage of participants
Arm/Group | 15 mg or MTD - Tirzepatide | 2.4 mg or MTD - Semaglutide
Number analyzed (Participants) | 318 | 318
Percentage of participants | 55.0 | 31.1

5. Secondary Outcome: Percentage of Participants Who Achieve ≥25% Body Weight Reduction
Description: Percentage of participants who achieved ≥25% body weight reduction (observed values) was reported.
Time Frame: Week 72
Population: All participants who received at least one dose of study drug and had evaluable data for this outcome.
Measure: Number; unit: Percentage of participants
Arm/Group | 15 mg or MTD - Tirzepatide | 2.4 mg or MTD - Semaglutide
Number analyzed (Participants) | 318 | 318
Percentage of participants | 36.5 | 18.6

6. Secondary Outcome: Change From Baseline in Waist Circumference in Centimeter
Description: Change from baseline in waist circumference in centimeter was reported. LS mean was determined using ANCOVA model with Baseline + Baseline BMI Group 1 + Sex + Pre diabetes status at randomization + Treatment (Type III sum of squares) as variables.
Time Frame: Baseline, Week 72
Population: All participants who received at least one dose of study drug and had evaluable data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: centimeters
Arm/Group | 15 mg or MTD - Tirzepatide | 2.4 mg or MTD - Semaglutide
Number analyzed (Participants) | 318 | 318
centimeters | -18.4 (0.61) | -13.0 (0.66)
Statistical Analysis 1: Comparison: 15 mg or MTD - Tirzepatide vs 2.4 mg or MTD - Semaglutide; Test type: Superiority; LS Mean Difference = -5.4, 95% CI 2-sided [-7.1 to -3.6]

7. Secondary Outcome: Percentage of Participants Who Achieve ≥30% Body Weight Reduction
Description: Percentage of participants who achieved ≥30% body weight reduction (observed values) was reported.
Time Frame: Week 72
Population: All participants who received at least one dose of study drug and had evaluable data for this outcome.
Measure: Number; unit: Percentage of participants
Arm/Group | 15 mg or MTD - Tirzepatide | 2.4 mg or MTD - Semaglutide
Number analyzed (Participants) | 318 | 318
Percentage of participants | 23.0 | 8.2

8. Secondary Outcome: Change From Baseline in Body Mass Index (BMI)
Description: Change from baseline in BMI was reported. LS mean was determined using Mixed Model Repeated Measures (MMRM) model using Baseline + Sex + Pre diabetes status at randomization + Treatment + Time + Treatment*Time(Type III sum of squares) as variables.
Time Frame: Baseline, Week 72
Population: All participants who received at least one dose of study drug and had evaluable data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: kilograms per meter square
Arm/Group | 15 mg or MTD - Tirzepatide | 2.4 mg or MTD - Semaglutide
Number analyzed (Participants) | 367 | 373
kilograms per meter square | -8.5 (0.24) | -6.0 (0.24)
Statistical Analysis 1: Comparison: 15 mg or MTD - Tirzepatide vs 2.4 mg or MTD - Semaglutide; Test type: Superiority; LS Mean Difference = -2.6, 95% CI 2-sided [-3.2 to -1.9]

9. Secondary Outcome: Percent Change From Baseline in Body Weight Comparing 15 mg Tirzepatide and 2.4 mg Semaglutide
Description: Percent change from baseline in body weight comparing 15mg of Tirzepatide and 2.4 mg Semaglutide was reported. The treatment effect for tirzepatide versus semaglutide for percent change in body weight was also evaluated assuming that participants had stayed on treatment and reached the highest dose of treatment. LS mean was determined by MMRM model using Baseline + Sex + Pre diabetes status at randomization + Baseline BMI Group 1 + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, Week 72
Population: All participants who received at least one dose of study drug and had evaluable data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | 15 mg or MTD - Tirzepatide | 2.4 mg or MTD - Semaglutide
Number analyzed (Participants) | 367 | 373
Percent change | -21.8 (0.60) | -15.4 (0.60)
Statistical Analysis 1: Comparison: 15 mg or MTD - Tirzepatide vs 2.4 mg or MTD - Semaglutide; Test type: Superiority; LS Mean Difference = -6.4, 95% CI 2-sided [-8.0 to -4.7]

ADVERSE EVENTS:
Time Frame: Baseline Up To 72 Weeks
Description: All randomized participants who received at least one dose of study drug. Gender specific events occurring only in male or female participants have had the number of participants at risk adjusted accordingly. Based on the planned safety analysis, adverse event analysis was planned as per the treatment regimen received.
Arm/Group | 15 mg or MTD - Tirzepatide | 2.4 mg or MTD - Semaglutide
All-Cause Mortality (participants affected / at risk) | 0/374 | 0/376
Serious Adverse Events (participants affected / at risk) | 18/374 | 13/376
Other Adverse Events (participants affected / at risk) | 255/374 | 267/376
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 15 mg or MTD - Tirzepatide (N=374) | 2.4 mg or MTD - Semaglutide (N=376)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Incarcerated hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Volvulus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 3 (3)
Gallbladder disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/242 (0) | 1/243 (1)
Benign fasciculation syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient global amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 15 mg or MTD - Tirzepatide (N=374) | 2.4 mg or MTD - Semaglutide (N=376)
Abdominal distension (Gastrointestinal disorders) | 27 (50) | 24 (29)
Abdominal pain (Gastrointestinal disorders) | 24 (31) | 26 (29)
Constipation (Gastrointestinal disorders) | 101 (179) | 107 (167)
Diarrhoea (Gastrointestinal disorders) | 88 (227) | 88 (212)
Dyspepsia (Gastrointestinal disorders) | 22 (31) | 28 (40)
Eructation (Gastrointestinal disorders) | 37 (47) | 29 (37)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 23 (34) | 40 (59)
Nausea (Gastrointestinal disorders) | 163 (561) | 167 (505)
Vomiting (Gastrointestinal disorders) | 56 (154) | 80 (218)
Fatigue (General disorders) | 39 (108) | 46 (72)
Injection site reaction (General disorders) | 32 (376) | 1 (1)
Covid-19 (Infections and infestations) | 51 (54) | 47 (48)
Nasopharyngitis (Infections and infestations) | 17 (20) | 23 (28)
Sinusitis (Infections and infestations) | 11 (14) | 21 (23)
Upper respiratory tract infection (Infections and infestations) | 32 (36) | 43 (49)
Decreased appetite (Metabolism and nutrition disorders) | 17 (17) | 19 (20)
Dizziness (Nervous system disorders) | 24 (30) | 18 (21)
Headache (Nervous system disorders) | 27 (43) | 27 (44)
Alopecia (Skin and subcutaneous tissue disorders) | 31 (31) | 23 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-08-24): https://cdn.clinicaltrials.gov/large-docs/30/NCT05822830/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-23): https://cdn.clinicaltrials.gov/large-docs/30/NCT05822830/SAP_001.pdf